CLINICAL TRIAL: NCT03649503
Title: The National Registry Study For the Real-world Patients With Parkinsonian Disorders in China (ForPDCN)
Brief Title: The National Registry Study For the Real-world Patients With Parkinsonian Disorders in China
Acronym: ForPDCN
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Tianjin Medical University General Hospital (Other); Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other); Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital of the Fourth Military Medical University (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Changshu Hospital of Traditional Chinese Medicine (Other); The Affiliated Hospital of Qingdao University (Other); Guangxi Ruikang Hospital (Other); Xi'an Central Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The First Hospital of Hebei Medical University (Other); Jieyang People's Hospital (Other); Luoyang Central Hospital (Other); Taian City Central Hospital (Other); Gansu Provincial Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Daqing Oil Field Hospital (Other); Fujian Provincial Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Taizhou Hospital (Other); Zhejiang Hospital (Other); The 101st Hospital of Chinese People's Liberation Army (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Dalian Medical University (Other); China-Japan Union Hospital, Jilin University (Other); Wuhan No.1 Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Northern Jiangsu People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Shanghai 5th People's Hospital (Other); Third People's Hospital, Huzhou City, Zhejiang Province, China (Other); Suzhou Municipal Hospital (Other); Ningbo No. 1 Hospital (Other); The First People's Hospital of Changzhou (Other); Affiliated Hospital of Jiangsu University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Fujian Medical University Union Hospital (Other); Shanghai Changzheng Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Jingjiang People's Hospital (Other); Qingdao Municipal Hospital (Other); Xi'an No.3 Hospital (Other Government); Lianyungang Hospital Affiliated Bengbu Medical College (Other); Jinzhou Medical University (Other); Shanghai 10th People's Hospital (Other); Huadong Hospital (Other); No. 102 Hospital of Chinese People's Liberation Army (Other); Shandong Provincial Hospital (Other Government); Anhui Provincial Hospital (Other Government); Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Jian Wang, Professor & Deputy Director, Department of Neurology, Huashan Hospital
Other Study IDs: KY2016-214
Record Dates: First submitted 2018-08-02; First posted 2018-08-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Parkinsonian Disorders
Keywords: Brain Health; Brain Research; parkinsonism; prospective cohort study; large sample size
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
The overall goal of this project is to identify, assess and longitudinally monitor subjects who are interested in participating in this study. Participants will enroll through a platform named PaWei, and provide informed consent prior to any study activities. PaWei will collect a variety of information, including participants' demographic information, overall health, family history of Parkinson's Disease, other clinical information (clinical drug use, drug efficacy, and comorbid disorders), mood status, sleep, diet, exercise, memory complaints, online cognitive tests, the Short-Form 8-Item Parkinson's Disease Questionnaire (PDQ-8), Movement Disorder Society-Unified Parkinson's Disease Rating Scale IB & II (MDS-UPDRS IB & II), Non-Motor Symptom Aassessment Scale for Parkinson's Disease (NMSS) , Hoehn and Yahr Scale, and other scales related to quality of life, etal---all through self-reported online questionnaires. Participants will also be asked to return to the PaWei every 3 months at regular intervals, to complete follow-up scales related to quality of life, and neuropsychological assessments, etal. Anyone with Parkinsonian Disorders is welcome to participate.

DETAILED DESCRIPTION:
In April 2017, the investigators launched a platform named PaWei which contains an iOS and Android smartphone application for patients and doctors. The platform connects patients, doctors and researchers by establishing communication and data transfer between the cloud platform and the mobile applications over the internet. The PaWei app is made available for free to download through the Apple App Store and Android Market. Through national outpatient service, advertisement and community outreach, potential participants will be directed to the PaWei APP. The overall goal of this project is to identify, assess and longitudinally monitor subjects who are interested in participating in this study. Participants will enroll through the PaWei APP, and provide informed consent prior to any study activities.

The PaWei APP will include:

1. Information about the National Registry Study (who is eligible to participate, the goals of the project and other relevant information about investigators and sponsors involved in the Initiative).
2. Frequently Asked Questions (FAQs) such as "How will my information be used?", "How will patient information be safeguarded?", "What information will be requested?", "How much time will be required for registration and testing?" will be addressed for participants.
3. General information about Parkinsonian Disorders.

The National Registry Study will be a large, online database of volunteers who are interested in participating in this study. Anyone with Parkinsonian Disorders is welcome to join the Registry.

1. Participants will provide their email address or telephone number and create an account and username with the Registry.
2. The Registry will send an automatic email or short message to the participant to verify their email address or telephone number.
3. Participants will read the online Information Sheet and will be asked to provide their consent by clicking either "I consent" or "I decline." Participants who decline to participate in the Registry will be not included in our study.
4. Participants who give their consent will be permitted to continue through the registration process, which includes completing a battery of questionnaires designed to obtain a general understanding of participants health, medical history wellbeing.
5. In addition to questionnaires, participants will be able to complete online scales related to quality of life, and cognitive assessments.
6. Participants will be given the option to elect a Caregiver and/or Study Partner (CASP) to enrich their study profile.
7. Video recordings: Participants are asked to perform finger tapping, hand movements, and walking in MDS-UPDRS III test after being instructed by the video example, and then to upload the videos to the PaWei APP. The severity of motor dysfunctions on those videos can be judged by clinicians, and be potentially quantified in the future by AI technology under development.
8. Data validation: (1) The quality control of raw data is the initial step of data analysis for any successful research. In PaWei platform, the investigators take a strategy of assessing the data quality by identifying poor-quality data, like incomplete data and illogical data based on the logistic verification about consistency of relevant questions. (2) Automated feedback loops are employed with this strategy to enable real-time detection of incomplete data or illogical data, which can be used to improve data collection quality.
9. Participants may be referred to other research studies and/or clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Anyone with Parkinsonian Disorders is welcome to join the Registry.

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Registry is a large, online database of volunteers who would like to participate in the research. Anyone with Parkinsonian Disorders is welcome to join the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Short-Form 8-Item Parkinson's Disease Questionnaire (PDQ-8) Score | Baseline, year 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and final visit (last study visit or early withdrawal visit, up to 10 years)
  The short-form 8-item Parkinson's disease Questionnaire (PDQ-8) is the most commonly used scale measuring health related quality of life (HRQoL) in PD patients. It includes 8 items, and each item has five options (never, occasionally, sometimes, often, always or cannot do at all). The total scores range from 0 (good health) to 32 (poor health). The change of PDQ-8 score is defined as the score collected at visit 4 (end of year 1), visit 8 (end of year 2), visit 12 (end of year 3), visit 16 (end of year 4), visit 20 (end of year 5), visit 24 (end of year 6), visit 28 (end of year 7), visit 32 (end of year 8), visit 36 (end of year 9), visit 40 (end of year 10), and final visit (last study visit or early withdrawal visit, up to 10 years) minus baseline score.
  Analysis Method: Mixed Model Repeated Measures (MMRM)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided